CLINICAL TRIAL: NCT02053688
Title: Evaluation Study on Corneal Lens for Vision Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FORSIGHT Vision3 (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CL001
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Astigmatic Correction Lens (Active Comparator): Nexis ACCL lenses vs commercial Toric Lenses
  Interventions: Device: Astigmatic Correction Lens (Nexis ACCL lenses)
- Toric Soft Contact Lenses (Active Comparator): commercial toric soft contact lenses
  Interventions: Device: Toric Soft Contact Lenses

INTERVENTIONS:
Device: Astigmatic Correction Lens (Nexis ACCL lenses) — Astigmatic refractive error correction
  Arms: Astigmatic Correction Lens
Device: Toric Soft Contact Lenses — astigmatism correction using toric optics
  Arms: Toric Soft Contact Lenses

SUMMARY:
The objective of this study is to evaluate the fitting and visual outcomes of Nexis Lens, made of silicone commonly used in the contact lens industry, on healthy eye with or without astigmatism.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with good corneal health
2. Age 18-65.
3. Patients able to understand the requirements of the study and willing to follow study instructions, to provide written informed consent to participate, and who agree to comply with all study requirements.
4. Best corrected visual acuity of 20/20 or better in the study eye/s

Exclusion Criteria:

1. Any other anterior segment abnormality.
2. No previous corneal procedures, including Laser Vision Correction.
3. Any abnormalities associated with the eye lids.
4. Clinically significant inflammation or infection within six (6) months prior to study.
5. Uncontrolled systemic disease (e.g., diabetes, hypertension, etc.) in the opinion of the Investigator.
6. Participation in any study involving an investigational drug or device within the past 30 calendar days, or ongoing participation in a study with an investigational material except studies using corneal lenses.
7. Intolerance or hypersensitivity to topical anesthetics, fluorescein, or components of the material.
8. Specifically known intolerance or hypersensitivity to contact lenses.
9. Any condition that, in the opinion of the investigator, would jeopardize the safety of the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 30 mins

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Tuan, OD, PhD, Principal Investigator — Nexisvision
Locations (6):
- United States (6):
  - Cliff Leong, Fremont, California
  - Sara Chiu, Fremont, California
  - John Michelsen, Livermore, California
  - Nexis Vision, Menlo Park, California
  - Nick Chan, San Mateo, California
  - Josephine Vo-Laurel, Stockton, California